CLINICAL TRIAL: NCT00006220
Title: Arsenic Trioxide Alone or With ATRA (Vesanoid) for Resistant Hematologic Malignancy
Brief Title: Arsenic Trioxide With or Without Tretinoin in Treating Patients With Hematologic Cancer That Has Not Responded to Previous Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study drug became commercially available.
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CDR0000068108; WU-99-0236; NCI-V00-1608
Record Dates: First submitted 2000-09-11; First posted 2004-05-20 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; previously treated myelodysplastic syndromes; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — Arsenic Trioxide; Tretinoin

ARMS (3):
- Phase I (Experimental): Starting dose of arsenic trioxide of 0.15 mg/kg/day
  Interventions: Drug: arsenic trioxide
- Phase II (Experimental): MTD of arsenic trioxide
  Interventions: Drug: arsenic trioxide
- Treatment Failure (Experimental): Arsenic trioxide and tretinoin
  Interventions: Drug: arsenic trioxide; Drug: tretinoin

INTERVENTIONS:
Drug: arsenic trioxide
Drug: tretinoin
  Arms: Treatment Failure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Tretinoin may help hematologic cancer cells develop into normal white blood cells.

PURPOSE: Phase I/II trial to study the effectiveness of arsenic trioxide with or without tretinoin in treating patients who have hematologic cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
This is a dose escalation and efficacy study of arsenic trioxide. In the efficacy study, patients are stratified according to diagnosis (acute myelogenous leukemia vs acute lymphocytic leukemia vs myelodysplastic syndrome vs multiple myeloma vs non-Hodgkin's lymphoma and Hodgkin's disease). Phase I: Patients receive arsenic trioxide IV over 2 hours daily for 28 days. Treatment repeats every 42-59 days in the absence of disease progression or unacceptable toxicity. Patients who achieve complete remission (CR) or partial remission (PR) receive up to 4 courses. Patients who fail to achieve CR or PR or who experience disease progression may receive arsenic trioxide and tretinoin daily for 28 days every 42-59 days for up to 7 courses. Patients who fail to achieve CR or PR or experience disease progression with arsenic trioxide and tretinoin are removed from study. Cohorts of 3-6 patients receive escalating doses of arsenic trioxide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Phase II: Patients receive the MTD of arsenic trioxide as in phase I for up to 7 courses. Patients who fail to achieve CR or PR after 3 courses or experience disease progression are either taken off study or treated with arsenic trioxide and tretinoin as in phase I. Patients are followed monthly for 6 months, and then every 3 months for 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients with any of the following diagnoses: Acute lymphocytic leukemia OR acute myeloid leukemia Failed to achieve complete remission (CR) with induction chemotherapy OR Relapsed within one year of initial CR OR Relapsed after autologous or allogeneic transplant OR Any subsequent relapse OR Refractory following relapse CR2 or more (phase I only) Blastic phase chronic myelogenous leukemia Prior therapy allowed Myelodysplastic syndrome, including the following: Refractory anemia with excess blasts (RAEB) OR RAEB in transformation (high intermediate or high risk only) Relapsed after transplant CR2 or more (phase I only) Non-Hodgkin's lymphoma OR Hodgkin's disease Newly diagnosed or in first relapse and failed to achieve CR or partial remission after induction or salvage chemotherapy OR Second or later relapse OR Relapsed after transplant No disease that can be encompassed in a standard radiation port No asymptomatic, minimally symptomatic, or low grade lymphoma Multiple myeloma Symptomatic, progressive, or recurrent disease after treatment with alkylating agents, high dose corticosteroids, or anthracyclines OR Relapsed following transplant Not eligible for autologous or allogeneic transplant A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 500/mm3* Platelet count at least 50,000/mm3* *Unless caused by marrow infiltration by tumor No congenital bleeding disorder Hepatic: Bilirubin less than 2 times upper limit of normal (ULN) SGOT less than 3 times ULN Renal: Creatinine clearance greater than 25 mL/min Cardiovascular: No myocardial infarction, stroke, or unstable angina within the past 12 months No uncompensated congestive heart failure Left ventricular ejection fraction at least 40% Other: No active infection HIV negative HTLV I/II negative Not pregnant Fertile patients must use effective contraception during and for 2 years following study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Prior hydroxyurea allowed Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics Surgery: Not specified Other: At least 3 weeks since prior antileukemic therapy (except leukapheresis)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1999-06; Primary Completion 2000-11 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) | 28 days
Likelihood of complete (CR) or partial (PR) response following therapy | 6 months

SECONDARY OUTCOMES:
Explore the pharmacokinetics of arsenic trioxide alone and in combination with ATRA
Evaluate acute and chronic toxicities of arsenic trioxide alone and in combination with ATRA.
Determine the effects of arsenic trioxide alone and combined with ATRA on bcl-2, pml, and class I antigen expression and on apoptosis. Determine the effects of arsenic trioxide on T and B cell number and function
  Only when patients are circulating tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Randy A. Brown, MD, Study Chair — Washington University Siteman Cancer Center
Locations (1):
- Washington University Barnard Cancer Center, St Louis, Missouri, United States